CLINICAL TRIAL: NCT06287112
Title: Efficacy of ETGBD Parallel Insertion With Fully Covered Self-expandable Metal Stent for Preventing Acute Cholecystitis in Patients With Low Cystic Duct Insertion
Brief Title: Prevention of Acute Cholecystitis With ETGBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyun Paik, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PAC-ETGBD
Record Dates: First submitted 2024-02-20; First posted 2024-02-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Biliary Obstruction; Acute Cholecystitis
Keywords: Malignant biliary obstruction; Fully covered self expandable metal stent; Endoscopic transpapillary gallbladder drainage; Preventive Effect; Acute cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAC-ETGBD (Prevention of Acute Cholecystitis with ETGBD) (Experimental)
  Interventions: Device: Endoscopic transpapillary gallbladder drainage (ETGBD)

INTERVENTIONS:
Device: Endoscopic transpapillary gallbladder drainage (ETGBD) — Fully covered self-Expandable metal stent with Endoscopic transpapillary gallbladder drainage (ETGBD) in patient with cystic duct low insertion

SUMMARY:
The goal of this clinical trial is to learn about Efficacy of the ETGBD parallel insertion with fully covered self-expandable metal stent for preventing acute cholecystitis in patients with low cystic duct insertion.

In this study, we hypothesized that endoscopic transpapillary gallbladder drainage (ETGBD) with parallel insertion of a fully covered self-expanding metal stent(FCSEMS) through an endoscopic biliary drainage tunnel is superior in preventing complications such as cholecystitis when the gallbladder ducts confluence within the distal third of the common bile duct. And we aimed to confirm its efficacy by comparing the frequency, severity, and rate of invasive additional procedures due to cholecystitis complications to provide evidence of clinical utility.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19 years of age or older
2. Patients requiring endoscopic retrograde cholangiography and drainage for therapeutic purposes.
3. Patients with imaging (CT, Cholangiogram) confirmed confluence of the cystic duct with the distal third of the common bile duct.
4. Patients who have voluntary informed consent to participate in the study.

Exclusion Criteria:

* Patients who have undergone percutaneous/surgical bile duct or gallbladder drainage prior to study enrollment.
* Patients with anatomic deformity of the upper gastrointestinal tract after gastric or hepatobiliary surgery
* Patients with concomitant gastric/duodenal obstruction
* Patients with confirmed or suspected cystic duct obstruction on imaging studies
* Patients with acute cholecystitis, acute pancreatitis
* Patients who underwent cholecystectomy
* Patients with a life expectancy of less than 3 months
* Patients who are otherwise unable to undergo endoscopic retrograde cholangiopancreatography

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of acute cholecystitis | 2 months from the date of stent placement
  Diagnosis of Acute cholecystitis will be based on the Tokyo Guidelines 2018

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hyun Paik, MD., PhD., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided